CLINICAL TRIAL: NCT06002061
Title: Exploration of Potential Airway Muscle Activation on Sleep-Disordered Breathing Events Using Air Pressure Maneuvers
Brief Title: Airway Muscle Activation on Sleep-disordered Breathing Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovaResp Technologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Muscle Activation
Record Dates: First submitted 2023-08-01; First posted 2023-08-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: This study has been designed as a single group study, in which recruited patients who suffer from obstructive sleep apnea (OSA) will undergo one sleep study that will evaluate the effectiveness of applying brief air pressure maneuvers in activating the upper airway muscles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle Activation (Experimental): Participants in this arm will receive intervention via application of brief air pressure maneuvers.
  Interventions: Device: NovaResp MAPR System

INTERVENTIONS:
Device: NovaResp MAPR System — Baseline measurements will be taken while the subject is awake. Genioglossus activity with maximal tongue protrusion will be measured as well as the response to 1 to 2 pressure routines. Once the subject is sleeping, the operator will observe the PSG recording and determine sleep stage and respiratory phase (inspiration, expiration, between breaths). Test routines will be performed for each sleep stage and each respiratory phase. If the operator notices an apnea occurring, one of the routines will be applied. When all manual tests are complete, an "automatic" mode will be engaged for the remainder of the night. During this mode, a previously developed and trialled AI model will be used to predict if an obstructive apnea is upcoming. The operator will input which routine to test, and the routine will be automatically applied when a prediction occurs. There will be a minimum of 60 seconds between pressure routine applications.

SUMMARY:
The standard for treatment for people suffering from obstructive sleep apnea (OSA) syndrome involves the use of Continuous, or Automatic Positive Airway Pressure (CPAP, APAP) machines, which work by delivering air via tubing and mask to a patient at pressures of up to 20cmH2O. This increased pressure is meant to stabilize the airway to reduce obstruction events. APAP machines are generally more effective and more comfortable for patients than CPAP machines because these devices automatically adjust pressure to treat an apnea. As a result of the high rate of patient dissatisfaction with conventional PAP therapy, alternative treatments for sleep apnea have been developed. One therapeutic target for OSA is stimulation of the genioglossus muscle, a phasic respiratory muscle important in maintaining upper airway patency.

Recently, it has been shown that genioglossus reflex responses can be achieved through the application of negative pressure pulses as well as changes in airway pressure. These studies focused on activating pressure-sensitive mechanoreceptors within the upper airway known to contribute to genioglossus activity. Together, these studies have demonstrated that both brief pulses of negative airway pressure and changes in airway pressure are capable of eliciting genioglossus reflex responses.

The goal of this interventional study is to evaluate the potential of airway muscle activation on sleep-disordered breathing during sleep therapy by applying brief maneuvers of air pressure using existing pressure and flow sensors in conventional CPAP machines.

DETAILED DESCRIPTION:
Patients recruited for the study will undergo one overnight study period which will take place at the sleep clinic (Sleep Disorders Clinic, QEII Abbie J. Lane Memorial Building). Treatment will be delivered using a positive airway pressure (PAP) device with an Investigational Testing Authorization (ITA) from Health Canada (HC). This medical device consists of a commercially available PAP device which has been integrated with a feature to communicate with a computer hosting the software via USB. The custom software has been developed to allow an operator to specify the pressure routine to be applied using a laptop computer, which then controls the CPAP and applies the routine.

The patient's personal PAP therapy settings will be transferred to this device so that the the only modified part of their therapy will be the brief pressure maneuvers. Standard PSG which typically consists of EEG, electrooculography, surface EMG, and electrocardiogram measurements as well as a submental needle EMG will be used to measure genioglossal activity. EMG needle insertion will be performed by an Otolaryngologist. Prior to insertion of the EMG needle, patients will be offered local anesthetic 1-2% lidocaine. Natus coated stainless steel wires (0.38 mm in diameter) will be inserted into the genioglossus muscle submentally using a 28-gauge TECA® Elite Disposable Monopolar Needle. Tegaderm tape will be used to adhere wires to the skin. Participants will be asked to perform tongue protrusions (pushing the tongue as hard and fast as possible against the top two incisor teeth) and several large swallows to confirm correct placement of the electrode and to measure maximal genioglossal activity. The brief air pressure maneuvers will be applied both before falling asleep and while asleep to compare muscle activation in awake and asleep conditions as described in the test plan below:

There are 3 stages to the test, described below.

Stage 1: Subject is awake. To begin, baseline measurements will be taken while the subject is awake. Genioglossus activity with maximal tongue protrusion will be measured as well as the response to 1 to 2 pressure routines.

Stage 2: Subject is asleep, manual control. Once the subject is sleeping, the operator will observe the PSG recording and determine sleep stage and respiratory phase (inspiration, expiration, between breaths). Each of the test routines will be performed for each sleep stage and each respiratory phase. If the operator notices an apnea occurring, one of the routines will be applied.

The shapes of the pressure routines are illustrated below, and the table corresponds to the test parameters for each test routine to be applied. If significant arousal is being caused as noted on the EEG, higher levels of pressure amplitudes of the routines may be aborted.

Stage 3: Subject is asleep, automatic control. When all manual tests are complete, an "automatic" mode will be engaged for the remainder of the night. During this mode, a previously developed and trialled AI model will be used to predict if an obstructive apnea is upcoming. The operator will input which routine to test, and the routine will be automatically applied when a prediction occurs. There will be a minimum of 60 seconds between pressure routine applications.

ELIGIBILITY:
Inclusion Criteria:

* No history of self-reported, uncontrolled, severe cardiovascular or neurological issues
* Must be diagnosed with OSA
* Must be between 18 and 70 years old. People over 70 are excluded from this study, as they are more likely to have co-morbidities that overlap with the exclusion criteria for the study.
* Must be able to comply with all study requirements as outlined in the consent form
* Must be able to understand English and be willing to provide written informed consent
* Must be willing to lend their personal PAP device for inspection so that their personal PAP therapy settings can be transferred to one of our CPAP devices that has been modified to include the NovaResp MAPR System. Their device will not be used or modified during the study.
* Moderate or worse OSA (baseline AHI > 15 events/hour)
* BMI < 35 kg/m2

Exclusion Criteria:

* Subjects actively using bi-level PAP or require oxygen therapy
* History of severe cardiovascular disease, including NYHA Class III or IV heart failure, CAD with angina, or MI/stroke within past 6 months.
* Subjects who are medically complicated or who are medically unstable (i.e., cancer, dementia, unstable cardiac or respiratory disease, or unstable psychiatric illness)
* Potential sleep apnea complications that in the opinion of the clinician may affect the health and safety of the participant
* Inability or unwillingness of individual to give written informed consent
* Neuromuscular disease, hypoglossal-nerve palsy, severe restrictive or obstructive pulmonary disease, moderate-to-severe pulmonary arterial hypertension, severe valvular heart disease, New York Heart Association class III or IV heart failure, recent myocardial infarction or severe cardiac arrhythmias (within the past 6 months), persistent uncontrolled hypertension despite medication use, active psychiatric disease, and coexisting non-respiratory sleep disorders that would confound functional sleep assessment.
* A body-mass index (BMI; the weight in kilograms divided by the square of the height in meters) of more than 35.
* Pregnancy or planning attempting to become pregnant.
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Evaluating level of activation through EMG | 8 hours
  Raw genioglossus EMG data collected from the submental needle EMG will be rectified and processed using a moving-time average window and expressed as a percentage (units: %) of maximal EMG, as determined by initial baseline measurements. The data will be assessed for muscle activity in the periods where pressure routines were applied and compared between different types of routines and periods without pressure routines. The percentage of maximal EMG will indicate to what level muscle activation has occurred. This value will display activation of the upper airway muscles in response to the brief air pressure maneuvers.
Evaluating decrease in AHI | 8 hours
  The apnea-hypopnea index will be obtained through Polysomnography (PSG) data, which are standard measures obtained in sleep studies. AHI is measured as the average number of Apnea and Hypopnea occurrences in an hour during sleep (units: events/hour). A reduced AHI will display that the brief pressure maneuvers were successful in activating the upper airway muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Clinic, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No